CLINICAL TRIAL: NCT00194311
Title: Human Papillomavirus (HPV) Infection in Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Other Study IDs: 801452; R01HD042100-15 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Papillomavirus Infections; Pregnancy Complications
Keywords: HPV; Pregnancy
MeSH Terms: conditions — Papillomavirus Infections; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- pregnancy complications: prospective cohort study is to determine if maternal infection with Human papillomavirus (HPV) is associated with pregnancy complications including spontaneous preterm delivery (sPTD), severe preeclampsia (PE) (as per current ACOG: American College of Obstetrics and Gynecology criteria), and intrauterine growth restriction (IUGR).

SUMMARY:
The purpose of this study is to determine if maternal infection with human papillomavirus (HPV) is associated with pregnancy complications including spontaneous preterm delivery (sPTD), severe preeclampsia (PE), and poor fetal growth.

ELIGIBILITY:
Inclusion Criteria:

* All women presenting for prenatal care at the Hospital of the University of Pennsylvania or affiliated clinics

Exclusion Criteria:

* Multiple gestations
* Medical conditions such as diabetes, chronic hypertension, renal disease
* Fetal malformations or chromosomal anomalies
* Fetal death

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 620 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Parry, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States